CLINICAL TRIAL: NCT03993197
Title: New Perioperative and Non-pharmacological Practices in Endometriosis at the Crossroad of Gynecology and Chronic Pain
Brief Title: Endometriosis and Pain
Acronym: EndoDOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL18_0474; 2018-A02599-46 (Other: ANSM)
Record Dates: First submitted 2019-06-05; First posted 2019-06-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pain; group management; quality of life
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients suffering from severe endometriosis and chronic pain (Experimental): Patients suffering from severe endometriosis and chronic pain that have been identified during a gynecological consultation (individual or during a multidisciplinary team meetings) or during a pain consultation on the same site of the Croix-Rousse Hospital and having signed a consent form
  Interventions: Behavioral: Psychological and corporal group management

INTERVENTIONS:
Behavioral: Psychological and corporal group management — After inclusion, patient will be divided into groups of 6 or 8 patients either in pre-operative or post-operative phase. Patient care will take place entirely in pre-operative or post-operative phase.
  Each group will benefit of six one hour and a half sessions.
  The frequency is established as follows:
  * First week a session of Body Strategy ©
  * Second week a psychological session with group of speech (Photolanguage ©).
  * Third week is a break Then the cycle currently described is repeated, for a total of 6 alternate sessions

SUMMARY:
Endometriosis is a condition affecting about 10% of childbearing age women. It can begin a few months to a few years after puberty. It causes abdominal and pelvic pain that can be extremely debilitating, affecting the quality of patients life by affecting sexuality and fertility. Psychological repercussions are very important and underestimated. Patient care focuses most often on the "organ pathology treatment ".

This study proposes to evaluate a multidisciplinary patient care by insisting on anatomo-physiological pain management, psychological and bodily, in the perioperative phase.

The main objective is to evaluate benefit of psychological and corporal group management on the overall quality of life of patients with severe endometriosis in terms of endometriotic damage and/or functional and painful repercussions, requiring surgery, before or after this study

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years
* Patients with deep endometriosis according to the CNGOF (collège national des Gynécologues et Obstétriciens Français) and/or chronic pain related to endometriosis according to doctor's evaluation and to the definitions of IASP (International Association for the Study of Pain) and HAS (French National Authority for Health) in treatment failure despite appropriate medical or surgical management of endometriosis
* Patients with social security
* Patients willing to come to all study visits
* Patients who signed their informed consent

Exclusion Criteria:

* Patients unable to participate in group care:

  * Patients with social phobia assessed during the inclusion interview
  * Patients with psychiatric disorders of a psychotic nature: delirium, hallucination, incoherent thoughts
  * Patients with behavioral disorders of hetero-aggressive or self-aggressive type oPatients with a handicap that prevents them following the physical and psychological group sessions (speech disorders, hearing, visual or practical)
* Pregnant women
* Patients planning a change (stop, start) during the study of their psychological management in their current care path.
* Patients planning a change (stop, start) during the study of their treatment by non-medicinal techniques (auriculo-acupuncture, relaxation and self-hypnosis, transcutaneous neurostimulation by TENS)
* Patients suffering from other severe or chronic somatic diseases associated with endometriosis
* Patients with cognitive disorders
* Patients with analgesics addiction (psychoactive substances, morphine substances, etc.)
* Patients protected by law (under guardianship / trusteeship)
* Patients participating in another interventional research that may interfere with the protocol results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Evolution of Physical Component Score (PCS) assessed by the Medical Outcome Study Short Form -36 (MOS SF 36) scale | at 3 months
  The Physical Composite Score (PCS) is based on four physical dimensions of quality of life and involves 8 components (Physical Functioning, Role Physical, Bodily Pain,General Health, Vitality, Social Functioning,Mental Health and Emotional Role). The evolution of the PCS is measured between T0, start of care, and the end of care (at T0 + 3 months).
  The PCS score ranges from 0 to 100, a higher score being associated with a better quality of life.

SECONDARY OUTCOMES:
Evolution of pain: Visual Analogue Scale (VAS) | at 3 months
  Evolution of pain assessed by the Visual Analogue Scale (VAS) between the beginning (T0) and the end of patient care (T0 + 3 months), in different body areas (back - abdomen - pelvic area - others) The VAS allows patients to rate their pain in an objective and comparable measure. This allows a quantitative evaluation of intensity of pain and trace evolution of the symptomatology in the same subject.
  The VAS ranges from 0 to 10, 0 for no pain, 10 for maximum pain.
Evolution of overall pain: Visual Analogue Scale (VAS) | at 3 months
  Evolution of overall pain assessed by the Visual Analogue Scale (VAS) between the beginning (T0) and the end of patient care (T0 + 3 months) The VAS allows patients to rate their pain in an objective and comparable measure. This allows a quantitative evaluation of intensity of pain and trace evolution of the symptomatology in the same subject.
  The VAS ranges from 0 to 10, 0 for no pain, 10 for maximum pain.
Comparison of painful location on the body pain schema, before/after patient care | at 3 months
  Comparison of painful location (circle by the patient on the body schema) before (T0)/after patient care (T0 + 3 months).
  Since endometriosis is synonymous with chronic and specific chronic pain (dyspareunia, dyschesia, cystalgia, for example), the body pain schema is a complementary tool in measurements, where the patient precisely surrounds the painful location (localizations of pain) and their extensions on a body schema,
Comparison of area of pain on the body pain schema, before/after patient care | at 3 months
  Comparison of area of pain (circle by the patient on the body schema), before (T0)/after patient care (T0 + 3 months).
  Area of each pain location will be calculated using the Geocalcul.Plus software and will be compared between the beginning (T0) and the end of patient care (T0 + 3 months).
Comparison of results of the interview schedule | at 3 months
  Comparison of results of the interview schedule before (T0) and after patient care (T0 + 3 months). Interview schedule examines two dimensions :
  * Inter-individual: couple quality of life, sex life
  * Intra-individual: self-image/body image, infertility, emotional life, pre or postoperative felt
Evolution of analgesics consumption | at 3 months
  Consumption of analgesics at the end of the treatment (T0 + 3 months) is self-evaluated by the patient: decreased / stable / increased.
number of painful crises | at 3 months
  Number of painful crises is the comparison of seizures number in the month preceding treatment with seizures number in the last month of care
Evolution of the Vitality (VT) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Vitality (VT) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The VT score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Social Function (SF) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Social Function (SF) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The SF score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Mental Health (MH) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Mental Health (MH) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The MH score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Role Emotional (RE) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Role Emotional (RE) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The RE score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Physical Function (PF) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Physical Function (PF) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The PF score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Role Physical (RP) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Role Physical (RP) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The RP score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Bodily Pain (BP) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Bodily Pain (BP) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The BP score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the General Health (GH) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the General Health (GH) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The GH score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Health Thinking (HT) score of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Health Thinking (HT) score is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The HT score ranges from 0 to 100, a higher score being associated with a better quality of life.
Evolution of the Mental Component Score (MCS) of the MOS SF36 score, before/after treatment | at 3 months
  The evolution of the Mental Component Score (MCS) is determined by the MOS SF36 and measured between T0, start of care, and the end of care (at T0 + 3 months).
  The MCS ranges from 0 to 100, a higher score being associated with a better quality of life.
Evaluation of the patient compliance with group management sessions | at 3 months
  The collection of the number of group sessions performed by the patient allows assessment of patient compliance with group management sessions. This evaluation allows to assess potential biases due to poor compliance in the final analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Branche, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix Rousse Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: No